CLINICAL TRIAL: NCT04078906
Title: Does Parenteral Omega-3 Enriched Lipid Emulsion Reduce Incidence of Bronchopulmonary Dysplasia in Preterm Infants
Brief Title: SMOFlipid and Incidence of BPD in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Belal Alshaikh, Clinical Associate Professor of Pediatrics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB19-1088
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Very Low Birth Weight Infant; Bronchopulmonary Dysplasia
Keywords: Intravenous lipid emulsions; SMOF; Preterm Infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — SMOFlipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Conventional IVLE (Intralipid) from D0 at 1g/kg/day and increase by 1 g/kg daily till reaching 3 g/kg/day.
- Experimental group (Experimental): n3-LCPUFA enriched IVLE (SMOFlipid) from D0 at 1g/kg/day and increase by 1 g/kg daily till reaching 3 g/kg/day.
  Interventions: Other: n3-LCPUFA enriched Intravenous Lipid Emulsion

INTERVENTIONS:
Other: n3-LCPUFA enriched Intravenous Lipid Emulsion — To start from D0 at 1g/kg/day and increase by 1 g/kg daily till reaching 3 g/kg/day.
  Other Names: SMOFlipid
  Arms: Experimental group

SUMMARY:
Despite many advances in neonatal care in the recent years, bronchopulmonary dysplasia (BPD) continues to be the major cause of chronic lung morbidity in infants. The pathogenesis of BPD is multifactorial; however, inflammation remains the central pathway for all risk factors. Omega-3 long chain polyunsaturated fatty acids (n3-LCPUFAs) from fish oil are known to down-regulate systemic inflammation and oxidative stress. Currently used soybean-based fatty acid emulsion (Intralipid) contains mainly n6-LCPUFA. Intralipid does not maintain the in-utero balanced LCPUFA accretion. Furthermore, Intralipid has been shown to increase free radical production and to be associated with BPD. A new fatty acid emulsion enriched with n3-LCPUFA (SMOFlipid) improves the fatty acid profile and reduces pro-inflammatory agents.

This project aims primarily to study whether SMOFlipid can lower the rate of BPD in preterm infants compared to Intralipid.

DETAILED DESCRIPTION:
Intravenous lipid emulsions (IVLEs) is a core component of parenteral nutrition (PN) for providing calories and essential fatty acids. Until recently, Intralipid was the only available IVLE in North America. For a long time now, the use of Intralipid has been described to be associated with the development of BPD. Lack of sufficient lipid clearance in premature infants, augmented oxidative stress, deficiency of anti-inflammatory agents, and elevated pulmonary artery pressure have all shown to be potential causes for lung injury during the use of Intralipid.

Intralipid, made mainly of soybean oil, contains high amounts of n6-LCPUFA and low amounts of n3-LCPUFA. This results in prostaglandin synthesis favoring pro-inflammatory products and amplified oxidative stress. Current evidence indicates that well-balanced fatty acid supply is a crucial factor to reduce inflammation and oxidative stress. The concern about unbalanced n6:n3 ratio has led to the development of novel IVLEs, like SMOFlipid. SMOFlipid is composed of a mixture of soybean oil (30%), medium-chain triglycerides (MCT) (30%), olive oil (25%) and fish oil (15%). The combination of soybean oil and fish oil allows delivering balanced LCPUFA with n6:n3 ratio of 2.5:1 and provides sufficient amounts of the preformed n3-LCPUFA.

Interventions that improve n3-LCPUFA status have been shown to reduce pulmonary inflammation in animal models.

In humans, a study on extremely preterm infants has revealed a rapid decline in the n3-LCPUFA in the first week of life despite the use of Intralipid. Early restoration of an adequate ratio of LCPUFA to inhibit inflammation has gained interest in recent years. In an observational study by Skouroliakou et al., very low birth weight infants receiving SMOFlipid within 48 hours of birth and for at least 7 days had a lower incidence of BPD compared to the Intralipid control group. A recent systematic review and meta-analysis of 8 randomized control trials (7 compared SMOFlipid to Intralipid) was conducted to evaluate safety and efficacy of fish oil-enriched IVLEs in preterm infants. Infants who received fish oil-enriched IVLEs had significantly higher RBC membrane DHA and EPA. The meta-analysis showed no difference in all-cause mortality and overall complication rate in 238 infants receiving fish oil-enriched IVLEs. However, all the studies included in this meta-analysis were small. Furthermore, the studies focused mainly on laboratory findings, and did not aim to study effect on inflammation, oxidative stress or clinical outcomes. Studies from critically ill adults in intensive care units exhibited a reduction in the duration of hospitalization and ventilator days, a risk factor for lung injury, when using n3-LCPUFA enriched IVLEs.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <30 weeks and admitted to NICU at Foothills Medical Centre in the first 24 hours of life.
* Anticipated duration of PN for >7 days

Exclusion Criteria:

* Infants with congenital anomalies
* Infants with suspected inborn errors of metabolism or family history of inborn error of metabolism
* Perinatal asphyxia
* Evidence of congenital infection
* Primary biliary atresia

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of Bronchopulmonary Disease | 36 weeks corrected gestational age
  According to Child Health and Human Development with classification to mild, moderate and severe.
Fatty acid profile | First 3 weeks of life
  Determine serum fatty acids levels (μmol/L).
Pro-inflammatory cytokine response | First 3 weeks of life
  Compare pro-inflammatory cytokine levels (pg/mL)
Lipid peroxidation measure 1 | First 3 weeks of life
  Malondialdehyde (MDA, μmol/L) in blood
Lipid peroxidation measure 2 | First 3 weeks of life
  8-isoprostane levels (pg/mL) in blood

SECONDARY OUTCOMES:
Incidence of Cholestasis | Up to 36 weeks corrected gestational age or discharge
  Direct bilirubin more than 34 mmol/L
Weight gain velocity | Up to 36 weeks corrected gestational age or discharge
  Change in weight Z scores
Incidence of retinopathy of prematurity | Up to 36 weeks corrected gestational age or discharge
  Defined as stage 2 or higher according to the international classification or requiring treatment.
Incidence of moderate to severe neurodevelopmental disability | 18-22 months corrected gestational
  Defined by 1 or more of the following: moderate to severe motor impairment cerebral palsy (CP) or non-CP) with a GMFCS level ≥2, a BSID III cognitive score of <70, severe visual impairment (bilateral blindness with vision <20/200), or severe hearing impairment (permanent hearing loss that interferes with ability to understand or communicate with or without amplification).
Incidence of severe intraventricular hemorrhage (IVH) | Up to 36 weeks corrected gestational age or discharge
  Defined as grade 3 or higher

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No